CLINICAL TRIAL: NCT02014792
Title: Heart Rate Variability and Omega-3 Fatty Acid Status in Haemodialysis Patients: an Observational Pilot Study
Brief Title: Heart Rate Variability & Fatty Acid Status: Haemodialysis Patients
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Wendy Hall, Lecturer in Nutritional Sciences, King's College London
Other Study IDs: DNS9195677
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Chronic Kidney Disease
Keywords: Haemodialysis; Heart rate variability; n-3 PUFA
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood Plasma Washed and isolated red blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease, stage 5: Patients with stage 5 chronic kidney disease who have recently commenced haemodialysis treatment (within 6-10 weeks of starting treatment)

SUMMARY:
Studies suggest that dietary omega-3 fatty acids influence the extent to which the time interval between each heart beat varies (heart rate variability; HRV). Low HRV is associated with increased risk of sudden cardiac death (SCD). The purpose of this research is to investigate the relationship between 24 hour parameters of HRV and blood omega-3 fatty acid levels in patients who have recently commenced haemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 5 commencing haemodialysis,
* male or female,
* aged 40-80 y,
* written informed consent

Exclusion Criteria:

* history of chronic liver disease or neuropathy, infection or antibiotics within the last month.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending King's College Hospital and Guy's and St Thomas' Hospitals who have recently commenced haemodialysis treatment.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Erythrocyte eicsapentaenoic acid (EPA) + docosahexaenoic acid (DHA) content (% weight of total fatty acids) | 6-10 wk after commencing haemodialysis treatment
  Primary independent variable
24 hour heart rate variability (Triangular index and SDNN) | 6-10 weeks after commencing haemodialysis treatment
  Primary dependent variables. Triangular index and SDNN are indicators of overall variability

SECONDARY OUTCOMES:
24 h heart rate variability - longer phase parameters | 6-10 weeks after commencing haemodialysis
  Parameters of longer phase HRV: LF, VLF and SDANN
24 h heart rate variability - short-phase parameters | 6-10 weeks after commencing haemodialysis
  RMSSD, pNN50, HF
Nocturnal heart rate variability - all parameters | 6-10 weeks after commencing haemodialysis
  SDNN, Triangular index, LF, HF, VLF, SDANN, RMSSD, pNN50 calculating during nocturnal sleep-time
Plasma EPA+DHA content (% weight of total fatty acids) | 6-10 weeks after commencing haemodialysis6-10 weeks after commencing haemodialysis

OTHER OUTCOMES:
Complications of haemodialysis in first 6 weeks of starting treatment | 0-6 weeks after commencing haemodialysis
  Incidence of problems with dialysis access, inadequate urea reduction ratio, amount of excess oedematous fluid removed, serious adverse events
Background dietary intakes | 6-10 weeks after commencing haemodialysis
  Food frequency questionnaire
History of sleep apnoea | 6-10 weeks after commencing haemodialysis
  Epworth Sleepiness scale and Berlin questionnaire, plus relevant medical history
Weight | 6-10 weeks after commencing haemodialysis
Waist circumference | 6-10 weeks after commencing haemodialysis
12 month average blood pressure | 12 months prior to commencing haemodialysis treatment
Plasma lipids | 6-10 weeks after commencing haemodialysis
C-reactive protein | 6-10 weeks after commencing haemodialysis
Serum electrolytes | 6-10 weeks after commencing haemodialysis
  Sodium, potassium, calcium, phosphate

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Hall, PhD, Principal Investigator — King's College London; Iain Macdougall, FRCP, Study Chair — King's College Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - King's College London, London
  - King's College Hospital, London
  - Guy's and St Thomas' Hospital, London

REFERENCES:
- [Result] Pinto, A., MacLaughlin, H., Gray, R., & Hall, W. (2020). Heart rate variability and long chain n-3 PUFA in patients with chronic kidney disease commencing haemodialysis: A cross-sectional study. Proceedings of the Nutrition Society, 79(OCE2), E643. doi:10.1017/S0029665120005923
- See also: Abstract (13th European Nutrition Conference, FENS 2019, 15-18 October 2019, Malnutrition in an Obese World: European Perspectives) — http://www.cambridge.org/core/journals/proceedings-of-the-nutrition-society/article/heart-rate-variability-and-long-chain-n3-pufa-in-patients-with-chronic-kidney-disease-commencing-haemodialysis-a-crosssectional-study/8AFEC1E1F7F909C3E8840868C8E5BECA